CLINICAL TRIAL: NCT03243578
Title: Relationship Between Dietary Protein Intake and Fatal and Non-fatal Health Outcomes in 180,031 UK Biobank Participants
Brief Title: Relationship Between Dietary Protein Intake and Fatal and Non-fatal Health Outcomes
Status: Completed | Type: Observational
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Dr Stuart Gray, University of Glasgow
Other Study IDs: UKBProHealth
Record Dates: First submitted 2017-08-01; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Cardiovascular Diseases; Cancer; All-cause Mortality
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None as this is an observational study

SUMMARY:
The aim of the current study was to clarify the relationship between protein intake and health by using a very large, general population cohort study, UK Biobank, to study the associations between reported protein intake (expressed in g/day, g/kg/day and % of total energy intake) and three health outcomes (all-cause mortality, incidence CVD and cancer).

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* None

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment from the general population
Sampling Method: Probability Sample
Enrollment: 502628 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Mean of 7 years
  Date and cause of death were obtained from death certificates
CVD incidence | Mean of 6.1 years
  Date and cause of hospital admissions were identified via record linkage to Health Episode Statistics (HES) records for England and Wales and to the Scottish Morbidity Records (SMR01) for Scotland
cancer incidence | Mean of 6.1 years
  Data on cancer diagnoses for participants resident in England and Wales is provided to UK Biobank by the Medical Research Information Service, based at the National Health Service Information Centre (http://www.ic.nhs.uk/services/medical-research-informationservice). The Information Services Division (http://www.isdscotland.org/HealthTopics/Cancer/), which is a part of NHS Scotland, provides UK Biobank with the cancer data records for participants resident in Scotland.

IPD SHARING:
Plan to Share IPD: No
Whilst we will not make this data available it is available to all bona fide researchers via the UK Biobank